CLINICAL TRIAL: NCT02500849
Title: A Pilot Study to Evaluate the Feasibility, Safety and Engraftment of Zinc Finger Nuclease (ZFN) CCR5 Modified CD34+ Hematopoietic Stem/Progenitor Cells (SB-728mR-HSPC) in HIV-1 (R5) Infected Patients
Brief Title: Safety Study of Zinc Finger Nuclease CCR5-modified Hematopoietic Stem/Progenitor Cells in HIV-1 Infected Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: Sangamo Therapeutics (Industry); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14017
Record Dates: First submitted 2015-03-16; First posted 2015-07-17 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: HIV
Keywords: Gene therapy; Acquired Immunodeficiency Syndrome; HIV Infections; Retroviridae Infections; RNA Virus Infections; Virus Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Immunologic Deficiency Syndromes; Immune System Diseases; Busulfan; Pharmacologic Actions
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Retroviridae Infections; RNA Virus Infections; Virus Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Immunologic Deficiency Syndromes; Immune System Diseases | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1: (Experimental): target busulfan AUC levels: 8,000 µM*min (+/- 1,000)
  Interventions: Genetic: SB-728mR-HSPC Infusion 3 days following busulfan conditioning
- Cohort 2: (Experimental): busulfan AUC levels: 12,000 µM*min (+/- 1,000)
  Interventions: Genetic: SB-728mR-HSPC Infusion 3 days following busulfan conditioning

INTERVENTIONS:
Genetic: SB-728mR-HSPC Infusion 3 days following busulfan conditioning
  Other Names: busulfan

SUMMARY:
The purpose of the study is to evaluate the safety and feasibility of administering SB-728mR-HSPC after conditioning with busulfan.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the safety and feasibility of giving autologous SB-728mR-HSPC to HIV-1 (R5) infected patients who are being treated with cART and have undetectable virus but suboptimal CD4+ cell levels. To strengthen the possibility that CCR5-disrupted HSPCs engraft, patients will receive either a two- or three-day (Cohort 1 or Cohort 2) course of busulfan (dose targeting AUC of 4000 µM/day) before being infused with the genetically modified cells. At 9-12 months after SB-728mR-HSPC infusion, subjects who are aviremic with CD4 cell counts ≥600 cells/µL and have ≥1% CCR5-modified CD4 cells within the peripheral blood detected by pentamer PCR will undergo an ATI.

ELIGIBILITY:
Inclusion Criteria:

* Maximum age 75 years for cohort 1 and 65 years for cohort 2.
* HIV-1 R5 seropositive with no evidence of CXCR4-tropic virus.
* On cART with undetectable HIV-1 (<20 gc/ml HIV-1 RNA) for at least 12 months prior to screening evaluations.
* CD4+ T-cell counts ≥200 cells/µL and ≤750 cells/µL.
* No psychosocial conditions that would hinder study compliance and follow-up.
* Absence of clinically significant cardiomyopathy, congestive heart failure.

Secondary Eligibility Criteria (for registration):

* Complete G-CSF/Plerixafor mobilization of HSPC.
* Collect ≥7.5 x 10^6 CD34+ cells/kg in two aphereses.
* The SB-728mR-HSPC product passed all release testing

Exclusion Criteria:

* Use of AZT or maraviroc in the cART regimen.
* History of significant hematologic diseases such as leukemia, myelodysplasia, coagulopathy, and thromboembolism.
* Any AIDS-related opportunistic infection occurring within the past year such as tuberculosis, cryptococcosis and for which treatment has been unsuccessful as determined by the Principal Investigator.
* AIDS-related syndromes, infectious or otherwise, if perceived to cause excessive risk for morbidity post-HSPC infusion, as determined by the Principal Investigator.
* Patients with active HBV or HCV infection, i.e., HBV DNA and HCV RNA in blood, are excluded. Those with inactive, but past infection with HBV (positive HBV surface antigen or HBV surface antibody) or inactive HCV (positive HCV antibody), must have no cirrhosis, as determined by abdominal ultrasound with elastography.
* Active CMV retinitis or other active CMV-related organ dysfunction.
* CXCR4-tropic virus.
* Pregnant or nursing women.
* Any history of HIV-associated encephalopathy; dementia of any kind; seizures in the past 12 months; any perceived inability to directly provide informed consent.
* Participants may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy. Participation in prior investigational drug or medical device study within the previous 45 days.
* Current or history of immunomodulatory agent or steroid use.
* Prior therapy with HIV vaccine or gene therapy product.
* History of alcohol or substance abuse for the previous 12 months.
* Participants with active malignancies. However, participants with skin cancers, namely basal cell or squamous cell carcinoma, and malignancies treated with curative intent having no known active disease present for ≥2 years, may be eligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-03-10 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-08-24 (Estimated)

PRIMARY OUTCOMES:
Toxicity in subjects who received SB-728mR-HSPC after each busulfan dose level | 18 months

SECONDARY OUTCOMES:
Number of CD34+ HSPC collected, gene modified, and released throughout the manufacturing process | Approximately first 1-2 months on study

OTHER OUTCOMES:
Detection of CCR5 modified HSPC in bone marrow | Up to Month 12
Time to hematological recovery as measured by neutrophil and platelet engraftment time | Up to Year 5
Changes in CD4+ T-cell percentage after SB-728mR-HSPC infusion | Up to Year 5
Changes in CD4+ T-cell number after SB-728mR-HSPC infusion | Up to Year 5
Changes in CD4/CD8 ratio after SB-728mR-HSPC infusion | Up to Year 5
Detection of CCR5-modified PBMC in blood over time | Up to Year 5
HIV-1 RNA levels in plasma during the treatment interruption of antiretroviral medicines | ATI Day 0 and weeks 2, 4, 6, 8, 10, 12, 14, 16 and 28
Longitudinal changes of proviral DNA in PBMC | 18 months
Pharmacokinetic analysis of busulfan (AUC levels) | pre-busulfan and at 15, 30, 60, 180 and 240 min after end of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Y. Krishnan, MD, Principal Investigator — City of Hope Medical Center
Locations (5):
- United States (5):
  - City of Hope Medical Center, Duarte, California
  - UCLA CARE Center, Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - Quest Clinical Research, San Francisco, California
  - Circle CARE Center, LLC, Norwalk, Connecticut

REFERENCES:
- [Derived] DiGiusto DL, Cannon PM, Holmes MC, Li L, Rao A, Wang J, Lee G, Gregory PD, Kim KA, Hayward SB, Meyer K, Exline C, Lopez E, Henley J, Gonzalez N, Bedell V, Stan R, Zaia JA. Preclinical development and qualification of ZFN-mediated CCR5 disruption in human hematopoietic stem/progenitor cells. Mol Ther Methods Clin Dev. 2016 Nov 9;3:16067. doi: 10.1038/mtm.2016.67. eCollection 2016. PMID 27900346